CLINICAL TRIAL: NCT01429298
Title: Randomized Clinical Trial Comparing Intravenous Hydromorphone to Usual Care
Brief Title: Comparing Intravenous Hydromorphone to Usual Care
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Andrew Chang, MD, Principal Investigator, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MMC 09-11-346
Record Dates: First submitted 2011-09-02; First posted 2011-09-07 (Estimated); Results first posted 2018-04-20 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-04

CONDITIONS: Pain
Keywords: Acute; Pain; Emergency Department; Hydromorphone; Protocol
MeSH Terms: conditions — Pain; Emergencies | interventions — Hydromorphone; Analgesics, Opioid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hydromorphone (Experimental): 2 mg of IV dilaudid will be administered over 2-3 minutes as initial dose.
  Interventions: Drug: Hydromorphone
- Usual care (Active Comparator): The attending physician administers whatever IV opioid he/she deems appropriate in whatever dose he/she chooses for initial dosing
  Interventions: Drug: Usual care

INTERVENTIONS:
Drug: Hydromorphone — 2 mg IV hydromorphone over to 2-3 minutes
  Other Names: Dilaudid
  Arms: Hydromorphone
Drug: Usual care — Attending administers IV opioid of his choosing
  Other Names: Opioids
  Arms: Usual care

SUMMARY:
In this randomized controlled trial, 2 mg intravenous (IV) hydromorphone will be more efficacious than usual care (usual care is analgesic management according to the judgment of the attending physician caring for that patient) in emergency department (ED) patients aged 21-64 years. The primary efficacy outcomes are the proportion of patients in each arm who choose to forgo additional pain medication in 30 minutes of entry into the study and the change in numerical rating scale (NRS) pain scores from baseline to 30 minutes post baseline.

DETAILED DESCRIPTION:
Patients were randomized to the 2 mg IV hydromorphone group or usual care; allocation was generated with www.randomization.com, using sealed opaque envelopes opened in sequential order by the research assistants (RAs) immediately following enrollment. Patients randomly allocated to usual care received an initial dose of IV opioid; the type and dose of which was determined by the treating emergency physician (EP). Patients in the 2 mg hydromorphone group were allocated to receive 2 mg IV hydromorphone, administered slowly over 2 to 3 minutes. All patients were placed on 2 L O2 by nasal cannula. Subjects were blinded to the treatment they were assigned. At 30 minutes, both groups were asked the following scripted question: "Do you want more pain medication?" Patients in either group who answered or otherwise indicated "yes" had their treating attending physician notified, who then decided on further pain management. Those who answered or otherwise indicated "no" did not receive additional analgesic at that time. Attending physicians were thus able to treat patients' pain in any manner they deemed fit once this primary study endpoint was reached. In addition to acquisition of the primary endpoint, patients were also asked to rate their pain on a previously validated and reproducible standard verbal NRS ranging from 0 ("no pain") through 10 ("worst pain possible") at 15, 30, 45, 60, 90, and 120 minutes following administration of the initial opioid dose at time 0. For safety reasons, patients were monitored for a total of 120 minutes (i.e., 90 minutes past the primary study endpoint) to determine adverse effects. Systolic blood pressure, heart rate, oxygen saturation, nausea, vomiting, and pruritus were assessed at baseline and at 15, 30, 45, 60, 90, and 120 minutes after initial administration of opioid. Patients who experienced oxygen desaturation (defined as < 95%) were gently aroused if sleeping, asked to take several deep breaths, and repositioned into a sitting position if they had been in a reclined position. Nasal cannula oxygen was also increased to 4 L, and the treating attending physician was notified. Subsequent management, including the use of naloxone, was per the treating attending physician's discretion.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 21 years and less than 65 years: This is a study of non-elderly adult patients.
2. Pain with onset within 7 days: Pain within seven days is the definition of acute pain that has been used in ED literature.
3. ED attending physician's judgment that patient's pain warrants IV opioids: The factors that influence the decision to use parenteral opioids are complex. An approach that is commonly taken to address the issue of patient selection in drug trials is to use a specific condition (e.g., renal colic) that would generally be thought to be appropriately treated with an opioid analgesic, thereby eliminating individual judgment about eligibility for the study. However in order to maximize the external validity of the role of opioids in the ED setting, the investigators decided to enroll patients with a variety of diagnoses, all with a complaint of acute pain. Opioids are not an appropriate treatment for all patients who present with a complaint of pain (e.g., gastroenteritis, migraine). Therefore, unless there is a restriction to patients with a specific diagnosis, either an extensive list of diagnoses and situations in which opioids are indicated must be specified, or clinical judgment needs to be used. The investigators have opted for the latter, since it most closely approximates the circumstances of clinical practice.

Exclusion Criteria:

1. Use of other opioids or tramadol within past 24 hours: to avoid introducing assembly bias related to recent opioid use, since this may affect baseline levels of pain and need for analgesics.
2. Prior adverse reaction to opioids.
3. Chronic pain syndrome: frequently recurrent or daily pain for at least 3 months results in modulation of pain perception which is thought to be due to down-regulation of pain receptors. Examples of chronic pain syndromes include sickle cell anemia, osteoarthritis, fibromyalgia, and peripheral neuropathies.
4. Alcohol intoxication: the presence of alcohol intoxication as judged by the treating physician may alter pain perception.
5. Systolic Blood Pressure <90 mm Hg: Opioids can produce peripheral vasodilation that may result in orthostatic hypotension.
6. Oxygen saturation < 95% on room air: For this study, oxygen saturation must be 95% or above on room air in order to be enrolled.
7. Use of monoamine oxidase (MAO) inhibitors in past 30 days: MAO inhibitors have been reported to intensify the effects of at least one opioid drug causing anxiety, confusion and significant respiratory depression or coma.
8. C02 measurement greater than 46: In accordance with standard protocol, three subsets of patients will have their CO2 measured using a handheld capnometer prior to enrollment in the study. If the CO2 measurement is greater than 46 then the patient will be excluded from the study. The 3 subsets are as follows:

   * All patients who have a history of chronic obstructive pulmonary disease (COPD)
   * All patients who report a history of asthma together with greater than a 20 pack-year smoking history
   * All patients reporting less than a 20 pack-year smoking history who are having an asthma exacerbation

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2010-03; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Montefiore Emergency Department, The Bronx, New York, United States

REFERENCES:
- [Derived] Chang AK, Bijur PE, Lupow JB, John Gallagher E. Randomized clinical trial of efficacy and safety of a single 2-mg intravenous dose of hydromorphone versus usual care in the management of acute pain. Acad Emerg Med. 2013 Feb;20(2):185-92. doi: 10.1111/acem.12071. PMID 23406078

RESULTS

PARTICIPANT FLOW:
Groups:
- Hydromorphone: 2 mg of IV dilaudid will be administered over 2-3 minutes as initial dose.
  2 mg IV hydromorphone: 2 mg IV hydromorphone over to 2-3 minutes
Period: Overall Study
Arm/Group | Hydromorphone | Usual Care
Started | 175 | 175
Given IV Opioids | 171 (4 never given IV opioids) | 169 (6 never given IV opioids)
Completed | 171 | 169
Not Completed | 4 | 6
Not completed — Protocol Violation | 4 | 6

BASELINE CHARACTERISTICS:
Population: The discrepancy between the number of patients who completed the study and the number of patients analyzed is due to: missing primary outcome data (4), enrolled twice (2), and received IV ketorolac prior to enrollment (9). These patients completed the study, but had unusable, duplicate, or unavailable data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydromorphone | Usual Care | Total
Number analyzed (Participants) | 164 | 161 | 325
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (12.2) | 41.2 (12.3) | 41.3 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 91 | 192
  Male | 63 | 70 | 133
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 113 | 103 | 216
  African American | 38 | 41 | 79
  White | 10 | 12 | 22
  Other | 3 | 5 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 164 | 161 | 325
Weight [Mean (Standard Deviation); unit: lbs] | 195.4 (39) | 201.4 (42.8) | 198.4 (41)
Location of Pain [Count of Participants; unit: Participants]
  Abdomen | 101 | 110 | 211
  Other | 63 | 51 | 114
Pain Intensity [Count of Participants; unit: Participants] — Pain intensity is measured on the numerical rating scale (NRS) from 0 ("no pain") to 10 ("worst pain imaginable").
  Participants
    Score of 3-7 | 19 | 21 | 40
    Score of 8 | 22 | 22 | 44
    Score of 9 | 20 | 15 | 35
    Score of 10 | 103 | 103 | 206
Nauseated or vomited before receiving opioids in the ED [Count of Participants; unit: Participants]
  Yes | 96 | 99 | 195
  No | 67 | 62 | 129
  Unknown | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Declined Additional Medication at 30 Minutes
Description: Amount of patients who choose to forgo additional pain medication at 30 minutes post-baseline when asked the question, "Do you want more pain medication?"
Time Frame: 30 minutes
Population: The discrepancy between the number of patients enrolled and randomized and the number of patients analyzed is due to: never given IV opioids (10), missing primary outcome data (4), enrolled twice (2), and received IV ketorolac prior to enrollment (9)
Measure: Count of Participants; unit: Participants
Arm/Group | Hydromorphone | Usual Care
Number analyzed (Participants) | 164 | 161
Participants | 127 | 106

2. Primary Outcome: Mean Change in Pain Intensity Score From Baseline to 30 Minutes
Description: Pain intensity is measured on the numerical rating scale (NRS) with scores ranging from 0 ("no pain") to 10 ("worst pain imaginable"). The change in NRS score is calculated by subtracting the score at 30 minutes post treatment from the score at baseline, before treatment. The average of these values was calculated.
Time Frame: 30 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hydromorphone | Usual Care
Number analyzed (Participants) | 164 | 161
units on a scale | 6.7 (2.9) | 5.6 (3.2)

3. Post Hoc Outcome: Number of Participants Who Achieved at Least 50% Decline in NRS Pain Score at 30 Minutes
Time Frame: 30 minutes
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hydromorphone | Usual Care
Number analyzed (Participants) | 164 | 161
Participants | 136 | 111

4. Post Hoc Outcome: Number of Patients Who Achieved Absolute Pain Intensity Score of 3 or Less at 30 Minutes
Description: Pain intensity is measured on the numerical rating scale (NRS) with scores ranging from 0 ("no pain") to 10 ("worst pain imaginable")
Time Frame: 30 minutes
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hydromorphone | Usual Care
Number analyzed (Participants) | 164 | 161
Participants | 114 | 90

5. Post Hoc Outcome: Number of Participants Who Reported no Pain or Mild Pain at 30 Minutes
Time Frame: 30 minutes
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Hydromorphone | Usual Care
Number analyzed (Participants) | 164 | 161
Participants | 122 | 95

ADVERSE EVENTS:
Time Frame: 30 minutes
Description: The discrepancy between the number of patients enrolled and randomized and the number of patients analyzed is due to: never given IV opioids (10), missing primary outcome data (4), enrolled twice (2), and received IV ketorolac prior to enrollment (9)
Arm/Group | Hydromorphone | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/164 | 0/161
Serious Adverse Events (participants affected / at risk) | 0/164 | 0/161
Other Adverse Events (participants affected / at risk) | 61/164 | 33/161
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Hydromorphone (N=164) | Usual Care (N=161)
Oxygen Saturation <95% (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Heart Rate <50 beats/min (Cardiac disorders) | 5 | 4
Systolic blood pressure <90 mmHg (Vascular disorders) | 3 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 30 | 14
Nausea (Gastrointestinal disorders) | 18/67 | 9/62 — excluding patients who were nauseated or vomiting prior to receiving opioids
Vomiting (Gastrointestinal disorders) | 5/67 | 3/62 — excluding patients who were nauseated or vomiting before perceiving opioids

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes